CLINICAL TRIAL: NCT07198854
Title: Analysis of Risk Factors Affecting Mesenchymal Stem Cells Efficacy in Hepatitis B Related Acute-on-chronic Liver Failure
Brief Title: Risk Factors Affecting MSC Efficacy in ACLF Patients
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Professor, Sun Yat-sen University
Other Study IDs: RISFAC-MSCs
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable- observational study — This is a retrospective cohort study and intervention is not applicable.

SUMMARY:
Mesenchymal stromal cells (MSCs) are potential therapy for many diseases, with the ability of tissue regeneration, repair and immunomodulation. Acute-on-chronic liver failure (ACLF) is a severe disease with high mortality. Previous studies showed that MSCs can improve the outcomes of Hepatitis B virus (HBV)-related ACLF patients. However, there are still some ACLF patients who have not benefited from MSC treatment. Thus, searching for risk factors affecting MSC efficacy in ACLF patients is of great significance for promotion of MSCs therapy.

This retrospective study will perform at a single center in southern China. Consecutive HBV related-ACLF patients treated with MSCs at the Third Affiliated Hospital of Sun Yat-sen University from January 2010 to October 2018 will be included. The clinical data including survival status, liver functions, complications et al. will be collected and analyzed, with the purpose of identifying the risk factors of HBV-related ACLF patients received MSCs injection and improving the efficacy of MSCs therapy furtherly.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute-on-chronic liver failure; Positive serum HBV surface antigen for more than 6 months; Received MSCs infusion more than one time.

Exclusion Criteria:

* Systemic or local malignancy; Hepatitis C virus infection; HIV infection or other immunodeficiency disease; Marked organ dysfunction (e.g., renal dysfunction); Pregnancy or lactation; Hyperthyroidism or other primary thyroid diseases; Incomplete data or lost to follow-up; Hospital stay < 1 day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBV related-ACLF patients treated with MSCs at the Third Affiliated Hospital of Sun Yat-sen University from January 2010 to October 2018.
Sampling Method: Probability Sample
Enrollment: 446 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Survival status | 90 days
  The survival status and survival time of the participants after receiving MSCs infusion will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Shi M, Zhang Z, Xu R, Lin H, Fu J, Zou Z, Zhang A, Shi J, Chen L, Lv S, He W, Geng H, Jin L, Liu Z, Wang FS. Human mesenchymal stem cell transfusion is safe and improves liver function in acute-on-chronic liver failure patients. Stem Cells Transl Med. 2012 Oct;1(10):725-31. doi: 10.5966/sctm.2012-0034. Epub 2012 Oct 11. PMID 23197664
- [Background] Lin BL, Chen JF, Qiu WH, Wang KW, Xie DY, Chen XY, Liu QL, Peng L, Li JG, Mei YY, Weng WZ, Peng YW, Cao HJ, Xie JQ, Xie SB, Xiang AP, Gao ZL. Allogeneic bone marrow-derived mesenchymal stromal cells for hepatitis B virus-related acute-on-chronic liver failure: A randomized controlled trial. Hepatology. 2017 Jul;66(1):209-219. doi: 10.1002/hep.29189. Epub 2017 May 27. PMID 28370357
- [Background] Sarin SK, Choudhury A, Sharma MK, Maiwall R, Al Mahtab M, Rahman S, Saigal S, Saraf N, Soin AS, Devarbhavi H, Kim DJ, Dhiman RK, Duseja A, Taneja S, Eapen CE, Goel A, Ning Q, Chen T, Ma K, Duan Z, Yu C, Treeprasertsuk S, Hamid SS, Butt AS, Jafri W, Shukla A, Saraswat V, Tan SS, Sood A, Midha V, Goyal O, Ghazinyan H, Arora A, Hu J, Sahu M, Rao PN, Lee GH, Lim SG, Lesmana LA, Lesmana CR, Shah S, Prasad VGM, Payawal DA, Abbas Z, Dokmeci AK, Sollano JD, Carpio G, Shresta A, Lau GK, Fazal Karim M, Shiha G, Gani R, Kalista KF, Yuen MF, Alam S, Khanna R, Sood V, Lal BB, Pamecha V, Jindal A, Rajan V, Arora V, Yokosuka O, Niriella MA, Li H, Qi X, Tanaka A, Mochida S, Chaudhuri DR, Gane E, Win KM, Chen WT, Rela M, Kapoor D, Rastogi A, Kale P, Rastogi A, Sharma CB, Bajpai M, Singh V, Premkumar M, Maharashi S, Olithselvan A, Philips CA, Srivastava A, Yachha SK, Wani ZA, Thapa BR, Saraya A, Shalimar, Kumar A, Wadhawan M, Gupta S, Madan K, Sakhuja P, Vij V, Sharma BC, Garg H, Garg V, Kalal C, Anand L, Vyas T, Mathur RP, Kumar G, Jain P, Pasupuleti SSR, Chawla YK, Chowdhury A, Alam S, Song DS, Yang JM, Yoon EL; APASL ACLF Research Consortium (AARC) for APASL ACLF working Party.. Acute-on-chronic liver failure: consensus recommendations of the Asian Pacific association for the study of the liver (APASL): an update. Hepatol Int. 2019 Jul;13(4):353-390. doi: 10.1007/s12072-019-09946-3. Epub 2019 Jun 6. PMID 31172417
- [Background] Joladarashi D, Kishore R. Mesenchymal Stromal Cell Exosomes in Cardiac Repair. Curr Cardiol Rep. 2022 Apr;24(4):405-417. doi: 10.1007/s11886-022-01660-1. Epub 2022 Jan 29. PMID 35092595
- [Background] Perico N, Remuzzi G, Griffin MD, Cockwell P, Maxwell AP, Casiraghi F, Rubis N, Peracchi T, Villa A, Todeschini M, Carrara F, Magee BA, Ruggenenti PL, Rota S, Cappelletti L, McInerney V, Griffin TP, Islam MN, Introna M, Pedrini O, Golay J, Finnerty AA, Smythe J, Fibbe WE, Elliman SJ, O'Brien T; NEPHSTROM Trial Consortium. Safety and Preliminary Efficacy of Mesenchymal Stromal Cell (ORBCEL-M) Therapy in Diabetic Kidney Disease: A Randomized Clinical Trial (NEPHSTROM). J Am Soc Nephrol. 2023 Oct 1;34(10):1733-1751. doi: 10.1681/ASN.0000000000000189. Epub 2023 Aug 10. PMID 37560967
- [Background] Xiang XN, Zhu SY, He HC, Yu X, Xu Y, He CQ. Mesenchymal stromal cell-based therapy for cartilage regeneration in knee osteoarthritis. Stem Cell Res Ther. 2022 Jan 10;13(1):14. doi: 10.1186/s13287-021-02689-9. PMID 35012666